CLINICAL TRIAL: NCT03269175
Title: BENEFIT 15 Long-term Follow-up Study of the BENEFIT and BENEFIT Follow-up Studies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19215; 2017-001176-31 (EudraCT Number)
Record Dates: First submitted 2017-08-09; First posted 2017-08-31 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Multiple Sclerosis
Keywords: Clinically Isolated Syndrome suggestive of Multiple Sclerosis or Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm 15 years ago (Other): This long term study does not imply current study medication. It looks at the status 15 years after the clinicial trial (BENEFIT)
  Interventions: Other: Brain MRI; Other: Blood sampling
- Placebo arm, offered treatment at MS diagnosis or at Month 24 (Other): This long term study does not imply current study medication. It looks at the status 15 years after the clinicial trial (BENEFIT)
  Interventions: Other: Brain MRI; Other: Blood sampling

INTERVENTIONS:
Other: Brain MRI — Brain MRI will be performed
Other: Blood sampling — Blood samples will be taken

SUMMARY:
The purpose of this study is to obtain long-term clinical data from patients approximately 15 years after their first clinical event, who participated in the former BENEFIT 304747 study and were treated at least once within that study.

This study will collect clinical information on the disease course, on disability, relapses, cognitive function over time, quality of life, depression, fatigue, resource use, and employment status. In addition, brain MRI is performed.

ELIGIBILITY:
Inclusion Criteria:

* All subjects who were treated at least once in BENEFIT study 304747 are eligible for inclusion in the BENEFIT 15 study

Exclusion Criteria:

* Subjects who, according to the investigator's judgment, have medical, psychiatric, or other conditions that compromise the subject's ability to understand the purpose of the study
* Suspected clinical instability or unpredictability of the clinical course during the study(e.g., due to previous surgery or acute stroke)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
Number of subjects with diagnosis of multiple sclerosis within fifteen years after Clinically-Isolated Syndrome (CIS) according to McDonald 2001 and 2010 criteria | Over 15 years since the subject´s first clinical event
Disease course since start of BENEFIT as assessed at the time of BENEFIT 15 | Over 15 years since the subject's first clinical event
Time to first relapse | Over 15 years since the subject´s first clinical event
Time to recurrent relapse | Over 15 years since the subject´s first clinical event
Annualized relapse rate | Over 15 years since the subject´s first clinical event
Time to conversion to Clinically-Definite Multiple Sclerosis (CDMS) | Over 15 years since the subject´s first clinical event
Time to conversion to Secondary Progressive Multiple Sclerosis (SPMS) | Over 15 years since the subject´s first clinical event
Expanded Disability Status Scale these scores (EDSS score) for disability assessed by the investigator during the neurological examination | 15 years after the subject´s first clinical event
Number of subjects with confirmed and sustained 1-point EDSS progression (Disability progression) | Over 15 years since the subject´s first clinical event
Number of subjects with confirmed 2.5-point EDSS progression (Disability progression) | Over 15 years since the subject´s first clinical event
Multiple Sclerosis Functional Composite (MSFC) score (Neurological status) | Over 15 years since the subject´s first clinical event
  MSFC: Multiple Sclerosis Functional Composite
Paced Auditory Serial Addition Test (PASAT-3) score (Cognitive function) | Over 15 years since the subject´s first clinical event
Time to use of ambulatory device | Over 15 years since the subject´s first clinical event
Time to dependence on ambulatory device | Over 15 years since the subject´s first clinical event
Time to use of wheelchair | Over 15 years since the subject´s first clinical event
Employment status (Standardized questions) | At one single visit, 15 years after the subject's first clinical event
  The current employment will be recorded
Multiple sclerosis impact on employment | At one single visit, 15 years after the subject's first clinical event
Resource use assessment questions: Help from family/regular ambulatory services | At one single visit, 15 years after the subject's first clinical event
Resource use assessment questions: Additional ambulatory services during relapse | At one single visit, 15 years after the subject's first clinical event
Resource use assessment questions: Adaptions (past 6 months) | At one single visit, 15 years after the subject's first clinical event

SECONDARY OUTCOMES:
Symbol Digit Modalities Test score (SDMT score) | At one single visit, 15 years after the subject's first clinical event
  SDMT: Symbol Digit Modalities Test, Cognitive test
  For sustained attention, concentration and information processing speed
Relation of SDMT and FSMC (Fatigue Scale for Motor and Cognitive Functions) | At one single visit, 15 years after the subject's first clinical event
Relation of mental processing speed and MRI parameters | At one single visit, 15 years after the subject's first clinical event
European Quality of life - 5 Dimensions Health-related Quality of life (EQ-5D HRQoL) score | Over 15 years since the subject´s first clinical event
  EQ-5D: European Quality of Life - 5 dimensions Questionnaire measuring health-related quality of life
European Quality of Life-5 Dimensions Visual Analog Scale (EQ-5D VAS) score | Over 15 years since the subject's first clinical event
Functional Assessment of Multiple Sclerosis (FAMS score) | Over 15 years since the subject´s first clinical event
  FAMS: Functional Assessment of Multiple Sclerosis
  Questionnaire measuring health-related quality of life
Fatigue Scale for Motor and Cognitive Functions (FSMC score) | At one single visit, 15 years after the subject's first clinical event
Center of Epidemiological Studies for Depression (CES-D) score | At one single visit, 15 years after the subject's first clinical event
Time to second line therapy | Over 15 years since the subject´s first clinical event
Time to first disease-modifying therapies (DMT) other than IFNB-1b | Over 15 years since the subject´s first clinical event

CONTACTS AND LOCATIONS:
Locations (61):
- Austria (2):
  - Medizinische Universität Graz, Graz, Styria
  - Landeskrankenhaus - Universitätskliniken Innsbruck, Innsbruck
- Belgium (4):
  - CU Saint-Luc/UZ St-Luc, Bruxelles - Brussel
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - CHU de Liège, Liège
- Canada (3):
  - Ottawa Hospital-General Campus, Ottawa, Ontario
  - CHUM - Hopital Hotel-Dieu, Montreal, Quebec
  - Montreal Neurological Hospital, Montreal, Quebec
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Ostrava, Ostrava-Poruba
  - Vseobecna fakultni nemocnice v Praze, Prague
- Amtssygehuset Glostrup, Glostrup Municipality, Denmark
- Finland (2):
  - Tampereen yliopistollinen sairaala, keskussairaala, Tampere
  - Terveystalo Turku, Turku
- France (5):
  - Hôpital Pellegrin - Bordeaux, Bordeaux
  - Hopital general, Dijon
  - Hopital Roger Salengro, Lille
  - Hôpital Pasteur - Nice, Nice
  - Hôpital Pontchaillou, Rennes
- Germany (10):
  - Klinikum der Universität München Grosshadern, München, Bavaria
  - Bezirksklinikum, Regensburg, Bavaria
  - Krankenhaus Hennigsdorf, Hennigsdorf, Brandenburg
  - Universitätsklinik Gießen und Marburg GmbH, Marburg, Hesse
  - Sana Klinikum Offenbach GmbH, Offenbach, Hesse
  - Universitätsmedizin der Georg-August-Universität Göttingen, Göttingen, Lower Saxony
  - Heinrich-Heine-Universität Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Städt. Krankenhaus Martha-Maria Halle-Dölau gGmbH, Halle, Saxony-Anhalt
  - HELIOS Klinikum Erfurt GmbH, Erfurt, Thuringia
  - Universitätsklinikum Charite zu Berlin, Berlin
- Hungary (4):
  - Peterfy Sandor utcai Korhaz - Rendelointezet, Budapest
  - Uzsoki Utcai Korhaz, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Szent-Gyorgyi Albert Orvostudomanyi Egyetem, Szeged
- Hadassah Hebrew University Hospital Ein Kerem, Jerusalem, Israel
- Italy (5):
  - Ospedale San Raffaele, Milan, Lombardy
  - IRCCS Ist Neurologico Nazionale C.Mondino, Pavia, Lombardy
  - ASST Valle Olona, Varese, Lombardy
  - A.O.U. San Luigi Gonzaga, Turin, Piedmont
  - A.O.U. Città della Salute e della Scienza di Torino, Torino, Tuscany
- Helse Bergen HF Haukeland universitetssjukehus, Bergen, Norway
- Poland (5):
  - 10 Wojskowy Szpital Kliniczny z Poliklinika SPZOZ, Bydgoszcz
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Szpital im. N. Barlickiego, Lodz
  - Samodzielny Publiczny Szpital Kliniczny nr 4, Lublin
  - Uniwersytecki Szpital Kliniczny im. J. Mikulicza-Radeckiego, Wroclaw
- Instituto Português de Oncologia Francisco Gentil - Coimbra, Coimbra, Portugal
- Spain (6):
  - Hospital Universitario Virgen de la Macarena, Seville, Andalusia
  - Ciutat Sanitària i Universitària de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Ciutat Sanitària i Universitaria de la Vall d'Hebron, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Regional de Málaga, Málaga
  - Hospital Universitari i Politècnic La Fe, Valencia
- Sahlgrenska Universitetssjukhuset, Gothenburg, Sweden
- Switzerland (2):
  - Universitätsspital Basel, Basel, Canton of Basel-City
  - Inselspital Universitätsspital Bern, Bern
- United Kingdom (4):
  - Royal Hallamshire Hospital, Sheffield, South Yorkshire
  - Aberdeen Royal Infirmary, Aberdeen
  - Ninewells Hospital, Dundee
  - Charing Cross Hospital, London

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/